CLINICAL TRIAL: NCT03440437
Title: A Phase 1/2, Open-Label, Study to Evaluate the Safety and Anti-Tumor Activity of FS118, a LAG-3/PD-L1 Bispecific Antibody, as a Monotherapy and in Combination With Paclitaxel, in Patients With Advanced Malignancies
Brief Title: A Phase 1/2 Study of FS118 in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: invoX Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FS118-17101
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-07

CONDITIONS: Advanced Cancer; Metastatic Cancer; Squamous Cell Carcinoma of Head and Neck
Keywords: FS118; Immuno-oncology; bispecific antibody; check-point inhibitor; dose escalation; cohort expansion; PK; PD; biomarker; LAG-3; PD-L1; SCCHN; F-star
MeSH Terms: conditions — Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FS118 weekly (Experimental): The initial cohorts will enroll sequentially as single-participant cohorts. If no DLT or ≥Grade 2 study drug related adverse event is observed, then dosing will proceed in a 3+3 design followed by an expansion cohort of participants with SCCHN and an expansion SCCHN cohort in combination with Paclitaxel.
  Interventions: Drug: FS118; Drug: Paclitaxel

INTERVENTIONS:
Drug: FS118 — Dosing of participants will occur intravenously (IV) weekly in 3-week treatment cycles until iCPD (i.e., immune confirmed progressive disease), unacceptable toxicity, or discontinuation.
Drug: Paclitaxel — Dosing on Days 1, 8 and 15 of each 28 day cycle in combination with FS118 given on days 1, 8, 15 and 22 of each 28 day cycle.

SUMMARY:
This study will be conducted in adult participants diagnosed with advanced tumors to characterize the safety, tolerability, pharmacokinetics (PK), and activity of FS118. This is a Phase 1/2, multi-center, open-label, multiple-dose, first-in-human study, designed to systematically assess safety and tolerability, to identify the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) for FS118 in participants with advanced tumors and to determine the efficacy of FS118 in participants with squamous cell carcinoma of the head and neck (SCCHN) as monotherapy and in combination with paclitaxel. In addition to safety, pharmacokinetics, pharmacodynamics, immunogenicity and efficacy will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Age ≥18 years;
* Participants with histologically confirmed, locally advanced, unresectable, or metastatic solid tumors that progressed while on or after PD-1/PD-L1 containing therapy;
* Measurable disease;
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1;
* Life expectancy estimated to be at least 3 months;
* Highly effective contraception;
* Willing and able to provide written informed consent.

Expansion cohort only:

* Histologically and/or cytologically confirmed recurrent/metastatic (R/M) SCCHN that is not amenable to curative therapy by surgery or radiation;
* Only 1 prior anti-PD-1 or anti-PD-L1 therapy and documented PD-L1 scoring ≥1% by combined positive score or tumor proportion score as part of their treatment;
* An anti-PD-1 or anti-PD-L1 treatment regimen must be the last prior therapy before study enrollment, following no more than 2 prior systemic regimens for R/M SCCHN;
* Acquired resistance to an anti-PD-1- or anti-PD-L1-containing therapy;
* The participant agrees to undergo a pre-treatment and on-treatment core or excisional biopsy and the biopsy procedure is not judged to be high risk by the Investigator.

Exclusion Criteria:

All participants:

* Participant is deemed at high risk of fatal outcome in case of COVID-19;
* Participants with a history of COVID-19 and have not provided a negative test for SARS CoV-2 infection within 28 days of the planned first dose date with FS118;
* Prior therapy: Received systemic anti-cancer therapy within 28 days or 5 half-lives, of the first dose of study drug, or prior treatment with a LAG-3 inhibitor;
* Participants with active or documented history of autoimmune disease;
* History of uncontrolled intercurrent illness;
* Known infections;
* Uncontrolled CNS metastases, primary CNS tumors, or solid tumors with CNS metastases as only measurable disease;
* Prior history of or active interstitial lung disease or pneumonitis, encephalitis, seizures, severe immune related adverse events with prior PD-1/PD-L1 containing treatments;
* Significant cardiac abnormalities;
* Significant laboratory abnormalities;
* Intolerance to the investigational product or its excipients, or any condition that would significantly impair and/or prohibit the participants's participation in the study, as per the Investigator's judgment.

Expansion cohort only:

* Participant has nasopharynx or thyroid primary tumor site;
* History of severe immune-related toxicity during the prior treatment with checkpoint inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Dose escalation: Incidence of Treatment Emergent Adverse Events (Safety and Tolerability) | 12 months
  Incidence, severity and duration of adverse events will be assessed by CTCAEv4.03
Dose escalation: Serum Concentration vs time profile of FS118 | 7 months
  Blood samples for serum PK analysis will be obtained (concentrations measured in mcg/mL)
Dose escalation: Maximum Serum Concentration of FS118 | 7 months
  Blood samples for serum PK analysis will be obtained (Cmax measured in mcg/mL)
Dose escalation: Time to reach maximum serum concentration (Tmax) of FS118 | 7 months
  Blood samples for serum PK analysis will be obtained (Tmax measured in hours)
Dose escalation: Trough serum concentration (Ctrough) of FS118 prior to the next dose | 7 months
  Blood samples for serum PK analysis will be obtained (Ctrough measured in mcg/mL)
Dose escalation: Area under the serum FS118 concentration vs time Curve (AUC) | 7 months
  Blood samples for serum PK analysis will be obtained (AUC measured in d.mcg/mL)
Dose escalation: Systemic Clearance (CL) of FS118 | 7 months
  Blood samples for serum PK analysis will be obtained (CL measured in mL/day)
Expansion cohort: Disease control rate as assessed by RECIST 1.1 in evaluable participants with PD-L1 and LAG-3 positive SCCHN | 24 weeks
  Assessed by RECIST 1.1
Expansion cohort (FS118 + paclitaxel): Incidence of Treatment Emergent Adverse Events (safety and Tolerability) Incidence, severity and duration of adverse events | 12 months
  Assessed by CTCAE v 5.0

SECONDARY OUTCOMES:
Dose escalation: Disease Response as assessed by RECIST 1.1 and iRECIST | 7 months
  Assessed by RECIST 1.1 and iRECIST
Dose escalation and expansion cohort of FS118 + paclitaxel | 7 months
  Incidence of FS118 immunogenicity will include ADA detection and analysis (incidence measured in titre)
Expansion cohort: Disease Response as assessed by RECIST 1.1 and iRECIST in all SCCHN participants | 24 months
  Assessed by RECIST 1.1 and iRECIST
Expansion cohort: Incidence of Treatment Emergent Adverse Events (Safety and Tolerability) | 12 months
  Incidence, severity and duration of adverse events will be assessed by CTCAEv4.03
Expansion cohort: Maximum Serum Concentration of FS118 | 7 months
  Blood samples for serum PK analysis will be obtained (Cmax measured in mcg/mL)
Expansion cohort: Time to reach maximum serum concentration (Tmax) of FS118 | 7 months
  Blood samples for serum PK analysis will be obtained (Tmax measured in hours)
Expansion cohort: Trough serum concentration (Ctrough) of FS118 prior to the next dose | 7 months
  Blood samples for serum PK analysis will be obtained (Ctrough measured in mcg/mL)
Expansion cohort: Area under the serum FS118 concentration vs time Curve (AUC) | 7 months
  Blood samples for serum PK analysis will be obtained (AUC measured in d.mcg/mL)
Expansion cohort: Systemic Clearance (CL) of FS118 | 7 months
  Blood samples for serum PK analysis will be obtained (CL measured in mL/day)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory Healthcare, Atlanta, Georgia
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- France (5):
  - CHU Bordeaux, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Lyon Berard, Lyon
  - La Timone, Marseille
  - Centre Antoine Lacassagne, Nice

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yap TA, LoRusso PM, Wong DJ, Hu-Lieskovan S, Papadopoulos KP, Holz JB, Grabowska U, Gradinaru C, Leung KM, Marshall S, Reader CS, Russell R, Sainson RCA, Seal CJ, Shepherd CJ, Germaschewski F, Gliddon D, Stern O, Young L, Brewis N, Kayitalire L, Morrow M. A Phase 1 First-in-Human Study of FS118, a Tetravalent Bispecific Antibody Targeting LAG-3 and PD-L1 in Patients with Advanced Cancer and PD-L1 Resistance. Clin Cancer Res. 2023 Mar 1;29(5):888-898. doi: 10.1158/1078-0432.CCR-22-1449. PMID 36342102